CLINICAL TRIAL: NCT01066026
Title: Double-blind, Randomized and Controlled Clinical Trial to Compare Safety and Efficacy of a Metallic Cannula vs a Standard Needle for the Injection of Hyaluronic Acid Gel Dermal Filler (Restylane®) to Treat Nasolabial Folds
Brief Title: Safety and Efficacy of a Metallic Cannula Versus A Standard Needle for Soft Tissue Augmentation of the Nasolabial Folds
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hexsel Dermatology Clinic (Other)
Responsible Party: Principal Investigator, Doris Hexsel, MD, Hexsel Dermatology Clinic
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 08-CBED08-02
Record Dates: First submitted 2010-01-26; First posted 2010-02-10 (Estimated); Results first posted 2020-09-09 (Actual); Last update posted 2020-10-01 (Actual); Status verified 2020-09

CONDITIONS: Wrinkles
Keywords: metallic cannula; Hyaluronic acid
MeSH Terms: interventions — Hyaluronic Acid; Restylane

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Metallic cannula (Experimental): Nasolabial Fold with metallic cannula and hyaluronic acid injected. hyaluronic acid with metallic cannula or standard needle. Hyaluronic acid injected with the new tool
  Interventions: Procedure: hyaluronic acid with metallic cannula or standard needle.; Drug: Hyaluronic acid injected with the new tool.
- Standard needle (Active Comparator): Nasolabial Fold with standard needle and hyaluronic acid injected. hyaluronic acid with metallic cannula or standard needle.
  Interventions: Procedure: hyaluronic acid with metallic cannula or standard needle.

INTERVENTIONS:
Procedure: hyaluronic acid with metallic cannula or standard needle. — The sides of injection were randomized and both the subject and the evaluator were blind to it. The injections were performed according through two different devices:
  * In one of the sides, the hyaluronic acid (Restylane®) was injected in its conventional pharmaceutical presentation, with a standard needle which is part of the product's kit;
  * In the other side, the hyaluronic acid (Restylane®) was injected through a metallic cannula, which replaced the needle of the product's kit.
  Local analgesia was provided for both applications: topical analgesics 4% Lidocaine, for the application with the standard needle, and nerve block (Lidocaine 2%), where the application was performed with the metallic cannula.
  Other Names: Restylane
Drug: Hyaluronic acid injected with the new tool. — hyaluronic acid with metallic cannula.
  Other Names: Restylane
  Arms: Metallic cannula

SUMMARY:
The purpose of this study was to assess the safety and efficacy of a new metallic cannula to inject hyaluronic acid for dermal augmentation in the nasolabial folds compared to standard needle.

DETAILED DESCRIPTION:
This was a monocentric, prospective, randomized, phase II and double-blind study.

At the baseline visits, one investigator rated the severity of nasolabial folds on both left and right sides according to the mentioned scale, and a standard set of six photographs of the face (frontal, left side and right side for both the whole face and the lower face) were taken.

On the day of the injection, the main investigator injected 1ml of dermal filler - hyaluronic acid (Restylane®, Q-Med, Uppsala, Sweden) - for each subject. The injected amount was 0,5ml for the right nasolabial fold and 0,5ml for the left nasolabial fold. The sides will be randomized.

ELIGIBILITY:
Inclusion Criteria:

* Subjects agreeing to take part of the study, after being fully informed of the purpose and the nature of the investigation and after having signed the informed consent form
* Female subjects aged from 18 to 60
* Fitzpatrick phototype I to VI
* Presence of bilateral folds graded from 2 to 3 according to the Modified
* Fitzpatrick Wrinkle Scale
* Subjects that have never performed any treatment of nasolabial folds
* Female subjects of childbearing age that present a negative urine pregnancy test and are using an effective contraceptive method
* Subjects who will be available throughout the duration of the study
* Subjects with sufficient schooling and awareness to enable them to cooperate to the degree required by this protocol.

Exclusion Criteria:

* Use of systemic corticosteroids
* History of herpes in lip
* Inflammation or active infection in the area to be injected
* Any surgical treatment or cosmetic procedure in the area to be injected that interfere in study's outcomes
* Coagulation disorders or use of anticoagulants
* Previous hypersensitivity responses to Hyaluronic acid.
* Pregnant or women in breastfeeding, or women planning to become pregnant

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2009-07; Primary Completion 2010-01 (Actual); Study Completion 2010-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Doris Hesxel, MD, Principal Investigator — CBED
Locations (2):
- Brazil (2):
  - Brazilian Center for Studies in Dermatology, Porto Alegre, Rio Grande do Sul
  - Centro Brasileiro de Estudos em Dermatologia, Porto Alegre

RESULTS

PARTICIPANT FLOW:
Groups:
- Metallic Cannula: Standard needle and metallic cannula were used in the same patient, with split face.
Period: Overall Study
Arm/Group | Metallic Cannula
Started | 25 (Each patient was injected with hyaluronic acid in each nasolabial fold (total: 2 injections))
Completed | 23
Not Completed | 2

BASELINE CHARACTERISTICS:
Groups:
- Metallic Cannula and Standart Cannula: Nasolabial Folds received fullers with Metallic Cannula or with Standard Needle
Arm/Group | Metallic Cannula and Standart Cannula
Number analyzed (Participants) | 25
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 25
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 50 (7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25
  Male | 0
Region of Enrollment [Number; unit: participants]
  Brazil | 25

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Haematoma
Description: Number of participants with haematoma at each visit
Time Frame: Day 1; day 3; day 7; day 90
Measure: Count of Participants; unit: Participants
Groups:
- Metallic Cannula; Standard Needle: Split face; metallic cannula on one side of the face and standard needle on the contralateral side (same patient).
Arm/Group | Metallic Cannula | Standard Needle
Number analyzed (Participants) | 25 | 25
Participants
  Day 1 | 10 | 23
  Day 3 | 6 | 11
  Day 7 | 1 | 4
  Day 90 | 0 | 0
Statistical Analysis 1: Comparison: Metallic Cannula vs Standard Needle; Test type: Non-Inferiority or Equivalence — pilot study; p < 0.0001, McNemar; descritive variables = 50, 95% CI 2-sided [5 to 95] — 50 was the percentage of hematomas expected for standard needle group

2. Primary Outcome: Number of Participants With Erythema
Description: Number of participants with erythema at each visit
Time Frame: Day 1; day 3; day 7; day 90
Measure: Count of Participants; unit: Participants
Arm/Group | Metallic Cannula | Standard Needle
Number analyzed (Participants) | 25 | 25
Participants
  Day 1 | 22 | 25
  Day 3 | 0 | 1
  Day 7 | 0 | 0
  Day 90 | 0 | 0

3. Secondary Outcome: Modified Fitzpatrick Wrinkle Scale (MFWS)
Description: Class 0 - No visible wrinkles; continuous skin lines Class 0.5 - Very shallow yet visible wrinkles Class 1 - Fine wrinkles. Visible wrinkles and slight indentations Class 1.5 - Visible wrinkles and clear indentations,<1-mm wrinkle depth* Class 2 - Moderate wrinkles. Clearly visible wrinkles, 1- to 2-mm wrinkle depth* Class 2.5 - Prominent and visible wrinkles; 2- to 3-mm wrinkle depth* Class 3 - Deep wrinkles. Deep, furrowed wrinkle; *>3-mm wrinkle depth
Time Frame: Baseline and 90 days
Population: Per protocol analysis. 23 participants attended to visit "Day 90'.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Metallic Cannula | Standard Needle
Number analyzed (Participants) | 23 | 23
scores on a scale
  Baseline | 2.40 (0.37) | 2.40 (0.37)
  Day 90 | 1.57 (0.57) | 1.54 (0.56)

4. Secondary Outcome: Global Aesthetic Improvement Scale
Description: 1. Very much improved: Optimal cosmetic result for the implant in this patient
  2. Much improved: Marked improvement in appearance from the initial condition but not completely optimal for this patient; touch-up would slightly improve the result
  3 - Improved: Obvious improvement in appearance from the initial condition, but touch-up or retreatment is indicated
  4 - No change: Appearance essentially the same as the original condition
  5 - Worse: Appearance worse than the original condition
Time Frame: 90 days
Population: Per protocol analysis. 23 participants attended to visit "Day 90'.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Metallic Cannula | Standard Needle
Number analyzed (Participants) | 23 | 23
scores on a scale | 2 (0.6) | 2 (0.7)

ADVERSE EVENTS:
Time Frame: 3 months
Description: pain,
Groups:
- Metallic Cannula: Nasolabial Fold with Metallic Cannula
- Standard Needle: Nasolabial Fold with standard needle
Arm/Group | Metallic Cannula | Standard Needle
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/25
Other Adverse Events (participants affected / at risk) | 0/25 | 0/25

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No